CLINICAL TRIAL: NCT01116505
Title: Treatment of Screen-detected Celiac Disease in Adults
Brief Title: Treatment of Screen-detected Celiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Kalle Kurppa, M.D, Ph.D, Pediatrician, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R07122
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Endomysial antibodies; Gluten-free diet; Screen-detected; Asymptomatic; Bone mineral density
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gluten-containing diet (No Intervention)
- Active comparator, gluten-free diet (Active Comparator)
  Interventions: Dietary Supplement: Gluten-free diet

INTERVENTIONS:
Dietary Supplement: Gluten-free diet — gluten-containing cereals removed from diet
  Arms: Active comparator, gluten-free diet

SUMMARY:
The main purpose of this study is to evaluate the natural history of celiac disease in asymptomatic, screen-detected subjects having positive endomysial antibodies and the effects of an intervention with a gluten-free diet. The investigators hypothesize that these subjects may have decreased general health and benefit of the dietary treatment regardless of the small-bowel mucosal structure.

DETAILED DESCRIPTION:
Asymptomatic, endomysial-antibody positive adults will be randomized to either continue with a normal, gluten-containing diet or start an intervention with a gluten-free diet irrespective of the small-bowel mucosal morphology. Several celiac-disease associated histological, serological and clinical markers will be evaluated both at baseline and after one year on trial.

ELIGIBILITY:
Inclusion Criteria:

* Positive endomysial antibodies
* Adults

Exclusion Criteria:

* Previous celiac disease diagnosis
* Significant clinical symptoms
* Suspicion of any serious celiac disease-associated complication
* Suspected or diagnosed severe illness other than celiac disease
* Consuming oral corticosteroids or immune suppressants
* Marked laboratory abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Small-bowel mucosal morphology and inflammation | One year

SECONDARY OUTCOMES:
Endomysial antibodies | one year
Tissue transglutaminase antibodies | one year
Antibodies to deamidated gliadin | one year
Intestinal tissue transglutaminase-specific IgA deposits | one year
Bone mineral density | one year
Body composition | one year
Health-related quality of life | one year
Laboratory parameters | one year

CONTACTS AND LOCATIONS:
Overall Officials: Katri Kaukinen, MD, Principal Investigator — University of Tampere, Tampere University hospital
Locations (1):
- Pediatric Research Centre, Tampere University Hospital and University of Tampere, Tampere, Pirkanmaa, Finland

REFERENCES:
- [Derived] Kurppa K, Paavola A, Collin P, Sievanen H, Laurila K, Huhtala H, Saavalainen P, Maki M, Kaukinen K. Benefits of a gluten-free diet for asymptomatic patients with serologic markers of celiac disease. Gastroenterology. 2014 Sep;147(3):610-617.e1. doi: 10.1053/j.gastro.2014.05.003. Epub 2014 May 13. PMID 24837306